CLINICAL TRIAL: NCT01974362
Title: Monolithic Zirconia Full-Mouth Implant Supported Rehabilitation Behavior
Status: Recruiting | Type: Observational
Sponsor: Implantology Institute (Other)
Responsible Party: Sponsor
Other Study IDs: II-06
Record Dates: First submitted 2013-10-26; First posted 2013-11-01 (Estimated); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Endosseous Dental Implant Failure; Accident Caused by Broken Ceramic
Keywords: Monolithic Zirconia; Zirconia-Feldspathic zirconia; Dental Implants; Fracture; Chipping
MeSH Terms: conditions — Fractures, Bone | interventions — Dental Implants

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Monolithic Zirconia with Buccal Veneer (MZ): Patients that have a full-mouth (maxilla and/or mandible) dental implant supported rehabilitation restored with monolithic zirconia biomaterial with buccal veneers
  Interventions: Device: Dental Implant; Device: Monolithic Zirconia (MZ)
- Monolithic Zirconia full-contour (FCMZ): Patients that have a full-mouth (maxilla and/or mandible) dental implant supported rehabilitation restored with monolithic zirconia biomaterial full contour (without veneer)
  Interventions: Device: Dental Implant; Device: Monolithic Zirconia (FCMZ)
- Zirconia-Feldspathic (PVZ): Patients that have a full-mouth (maxilla and/or mandible) implant supported rehabilitation restored with zirconia substructure and feldspathic veneered biomaterial
  Interventions: Device: Dental Implant; Device: Zirconia-Feldspathic (PVZ)

INTERVENTIONS:
Device: Dental Implant — Place dental implants in both jaws (maxilla and mandible) according to manufacturer specifications
  Other Names: Dental Fixtures
Device: Monolithic Zirconia (MZ) — rehabilitation with monolithic zirconia implant-prosthesis with bucal feldspathic veneer
  Other Names: Prettau®, Zirkonzhan®
  Groups: Monolithic Zirconia with Buccal Veneer (MZ)
Device: Zirconia-Feldspathic (PVZ) — restore dental implants with a zirconia suprastructure and feldspathic veneers
  Other Names: Ice Ceramic ® Zirkonzhan®
  Groups: Zirconia-Feldspathic (PVZ)
Device: Monolithic Zirconia (FCMZ) — Full contour full arch zirconia rehabilitation
  Other Names: Prettau®, Zirkonzhan®
  Groups: Monolithic Zirconia full-contour (FCMZ)

SUMMARY:
In patients that did a full mouth implant supported rehabilitation does Cad/Cam Monolithic Zirconia compared to Cad/Cam Zirconia Suprastructure (zirconium oxide (Yttrium - partially stabilized with tetragonal polycrystalline structure) veneered with feldspathic ceramic, has less post-insertion complications after at least 1-Year follow-up ?

DETAILED DESCRIPTION:
Study the behavior of implant supported rehabilitations made from full-zirconium dioxide (monolithic with buccal veneer (MZ) or full contour monolithic (FCMZ) ) and zirconia veneered with feldspathic (PVZ) in full-mouth type of rehabilitations (maxilla and mandible).

In a private clinic we will record the behavior, regarding prosthodontic and biological complications in different groups (MZ vs FCMZ vs PVZ) after at least 1 year in function.

We will make calibration of the investigators for prosthodontic and biological assessement and accepting an inter-observer agreement (Kappa) of 0.9 for each parameter.

Recording will be made without the help of magnifying utilities such as magnifying glasses or optical microscopes.

ELIGIBILITY:
Inclusion Criteria:

* Maxilla and/or Mandible Implant full-mouth restoration
* Monolithic ceramic or zirconia-feldspathic restoration
* be at least 18 years of age;
* present no systemic or local absolute contraindications for endosseous implant placement;
* at least 1 Year Follow-up

Exclusion Criteria:

* the presence of any systemic disease or condition that could compromise postoperative healing or osseointegration.
* Not full mouth rehabilitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients from a dental office that did a full-mouth (bimaxillary - maxilla and/or mandible) implant-supported rehabilitation and made the final rehabilitation with either monolithic zirconia or in feldspathic-zirconia
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Total Amount of Chipping | at least 1-Year post-insertion
  measure the total number of ceramic fractures (chipping) visible at naked eye in both groups (monolithic and feldspathic) that happen from insertion (baseline) to last follow-up visit
  Primary outcomes are defined as survival and success rates of the final prosthesis.
  For evaluation of these outcomes, an analysis variable will be used (Mendez Caramês et al., 2016): if no alterations are present, the prosthesis will be recorded as "Alpha"
Number of Small Complications | at least 1-year post-insertion
  Measure the total amount of adverse events other than chipping, that made the patient come to the dental office, that happen from insertion (baseline) to last follow up visit
  It is determined that if the complication was solved in the dental chair is considered a Small complication/minor chipping - not requiring any intervention besides polishing or recontouring without the need for prosthesis retrieval-"Bravo" classification will be attributed
Number of Big Complications | at least 1-Year post Insertion
  Measure the total amount of adverse events other than chipping, that made the patient come to the dental office, that happen from insertion (baseline) to last follow up.
  It is determined that if the complication was solved in the dental laboratory is considered a big complication/major chipping - a "Charlie" classification will indicate the occurrence of major chipping, need for prosthesis retrieval and laboratory intervention;
Number of prosthesis failures | at least 1-year post insertion
  a "Delta" classification will be attributed when fracture of the framework is present, defining a non-surviving prosthesis

SECONDARY OUTCOMES:
Biological complications | at least 1-Year post insertion
  implant success rates will be evaluated; absence of persistent subjective complaints (pain, foreign body sensation, and/ or dysesthesia); absence of peri-implant infection with suppuration; absence of implant mobility; and absence of continuous radiolucency around the implant by previously established methods based on the clinical and radiographic examinations at the yearly visits

CONTACTS AND LOCATIONS:
Overall Officials: João Caramês, Phd, Study Director — Implantology Institute; Artur Simões, Msc, Principal Investigator — Implantology Institute; Duarte Marques, Msc, Study Director — Implantology Institute
Locations (1):
- Artur Simões, Lisbon, Portugal

REFERENCES:
- [Result] Carames J, Marques D, Malta Barbosa J, Moreira A, Crispim P, Chen A. Full-arch implant-supported rehabilitations: A prospective study comparing porcelain-veneered zirconia frameworks to monolithic zirconia. Clin Oral Implants Res. 2019 Jan;30(1):68-78. doi: 10.1111/clr.13393. Epub 2018 Dec 30. PMID 30521106